CLINICAL TRIAL: NCT01988363
Title: Ultrasound-guided Greater Occipital Nerve Injection at Novel Proximal Location: A Clinical Series
Brief Title: Greater Occipital Nerve Injection Study
Acronym: GON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew Pingree, Assistant Professor of Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-005836
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Occipital Neuralgia; Cervicogenic Headache
Keywords: greater occipital nerve; occipital neuralgia; cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GON injection at C2 location (Other): A 25 gauge, 2 inch spinal needle will be inserted into the symptomatic side after locating the GON via US at the level of C2. Subjects will receive an injection of 4 ml of injectate consisting of 1 ml of 2% Lidocaine, 3 mg betamethasone and 2.5 ml of 0.25% Bupivicaine to the greater occipital nerve at the novel, proximal C2 location.
  Interventions: Procedure: GON injection at C2 location

INTERVENTIONS:
Procedure: GON injection at C2 location — GON will be identified at the novel, proximal C2 location on the symptomatic side via ultrasound guidance. Prior to injection, an independent examiner will perform a sensory exam of the involved dermatome. A 25 gauge spinal needle will be inserted into the symptomatic side after locating the GON via ultrasound at the C2 level. Subjects will be injected with treatment medication. Thirty minutes after injection, an independent examiner will test for anesthesia over the desired dermatome. VAS will be assessed pre-injection, 30 post-injection, 2 weeks post-injection and 1 month post-injection. The 2 week and 1 month assessments will be conducted by telephone.

SUMMARY:
This study is designed to answer the question of whether injection of the greater occipital nerve at its proximal origin, near the C2 vertebrae, using ultrasound guidance is effective in improving pain in human subjects.

HYPOTHESES

1. Ultrasound (US) guided greater occipital nerve (GON) injections are effective at a novel, proximal C2 location in live, human subjects, measured by improvement in visual analog scale (VAS) pain scores pre-injection compared to VAS scores 30 minutes post-injection, 2-weeks post-injection, and 1-month post-injection .
2. Ultrasound (US) guided injection of the greater occipital nerve (GON) at a novel, C2 location is effective at improvement of both occipital neuralgia and cervicogenic headache demonstrated by improvement in visual analog scale (VAS) pain scores pre-injection compared to VAS scores 30 minutes post-injection, 2-weeks post-injection, and 1-month post-injection. We further hypothesize that the mean improvement in VAS scores at 1-month post injection will be greater than 2 units.
3. Ultrasound (US) guided injection of the greater occipital nerve (GON) at novel, proximal C2 location in live, human subjects appears safe.

DETAILED DESCRIPTION:
Patients must be referred to Pain Clinic for occipital nerve injection.

Patients are responsible for all clinical costs associated with the injection.

There is no remuneration offered for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be referred to the Pain Clinic for an occipital nerve injection.

* Must have Occipital Neuralgia and/or Cervicogenic Headache

Exclusion Criteria:

* Bilateral GON symptoms and/or cervicogenic headache symptoms
* History of cervical spine surgery/procedure or trauma in past 6 months that may have caused or contributed to the occipital pain or cervicogenic headache, excluding Occipital Nerve Blocks (ONB).
* Evidence of impaired sensation in the GON dermatome region
* Evidence of cranial defect/abnormality near target injection site
* Untreated cutaneous infection, systemic illness, or immunocompromised state
* History of bleeding tendency or use of anticoagulants
* History of adverse reaction to anesthetic agents or corticosteroids
* Occipital nerve block in past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Successful anesthesia of the GON | 30 minutes post-injection
  Demonstration of successful anesthesia post-injection in the dermatomal distribution of the greater occipital nerve following ultrasound guided injections at a novel, proximal C2 location in live, human subjects.

SECONDARY OUTCOMES:
Change in Pain Scores | 30 minutes, 2 weeks, 1 month post-injection
  Obtain preliminary evidence of the efficacy of ultrasound guided greater occipital nerve injections at a novel, proximal C2 location in live, human subjects as measured by visual analog scale (VAS) pain scores pre-injection compared to VAS scores 30 minutes post-injection, 2 weeks post-injection and 1 month post-injection.

OTHER OUTCOMES:
Description of ultrasound GON injection | during injection
  To describe ultrasound guided greater occipital nerve injections in live, human subjects at a novel, proximal C2 location previously validated in cadaveric human models. This will include measurement of the cross-sectional area (mm^2), circumference (mm), depth from skin (cm) of the GON (cm), and presence or abscence of a vascular structure as measured with Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Pingree, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States